CLINICAL TRIAL: NCT02478593
Title: Impact of Patient Education on Benzodiazepine Use in the Elderly
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient funding
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Charles MacLean, MD, Professor of Medicine, Primary Care Internal Medicine, Department of Medicine Associate Dean for Primary Care, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 00000485
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2019-04

CONDITIONS: Anxiety; Insomnia
Keywords: Education; Geriatric; Benzodiazepine; Prevalence
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Group to receive educational booklet regarding risk/benefits of Benzodiazepine.
  Interventions: Behavioral: Educational booklet
- Control group (No Intervention): Group to receive educational booklet regarding risk/benefits of exercise.

INTERVENTIONS:
Behavioral: Educational booklet — Participants in the intervention group will receive an 8-page booklet that includes a list of generic and brand benzodiazepine names, benzodiazepine medication knowledge test, information about the associated risks of benzodiazepine use, and a list of safe alternative to their potentially inappropriate medication, as well as a stepwise tapering method. Recommendations to discuss decreasing use of benzodiazepines with physicians as well as to consult physicians before stopping any medication are also advised in the booklet. Participants in the control group will receive a booklet, produced by the Centers for Disease Control and Prevention, containing information regarding the important of exercise for seniors.
  Arms: Experimental group

SUMMARY:
The overall goal of this research is to develop and test strategies to decrease potentially inappropriate medication use among the elderly.

DETAILED DESCRIPTION:
Specifically, the purpose of the study is to determine whether direct patient education is effective in decreasing benzodiazepine use in seniors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Full benefit members living in a SASH facility
* 60 years old or older
* Using at least 1 active short/medium/long acting benzodiazepine at time of recruitment

Exclusion Criteria:

* Inability to provide consent
* Inability to communicate in English
* Diagnosis of severe mental illness, dementia, seizure disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06 (Estimated); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Benzodiazepine or non-benzodiazepine hypnotic medication use | Baseline and 6 months post-intervention
  Proportion of subjects using benzodiazepine or non-benzodiazepine hypnotic medication (such as zolpidem)

SECONDARY OUTCOMES:
Patient attempt to discontinuing benzodiazepine | 1 month and 6 months post-intervention
  Novel patient reported measure regarding attempts to discontinue medication
Patient knowledge regarding benzodiazepines | Baseline and 6 months post-intervention
  Novel patient reported measure regarding knowledge of the potential risks and benefits of benzodiazepines
Belief about Medicines Questionnaire (BMQ) | Baseline and 6 months post-intervention
  This is a validated instrument assessing patient beliefs regarding medication efficacy and safety

CONTACTS AND LOCATIONS:
Overall Officials: Charles MacLean, MD, Principal Investigator — University of Vermont

REFERENCES:
- [Result] Simon GE, Ludman EJ. Outcome of new benzodiazepine prescriptions to older adults in primary care. Gen Hosp Psychiatry. 2006 Sep-Oct;28(5):374-8. doi: 10.1016/j.genhosppsych.2006.05.008. PMID 16950371
- [Result] Charlesworth CJ, Smit E, Lee DS, Alramadhan F, Odden MC. Polypharmacy Among Adults Aged 65 Years and Older in the United States: 1988-2010. J Gerontol A Biol Sci Med Sci. 2015 Aug;70(8):989-95. doi: 10.1093/gerona/glv013. Epub 2015 Mar 1. PMID 25733718
- [Result] Weng MC, Tsai CF, Sheu KL, Lee YT, Lee HC, Tzeng SL, Ueng KC, Chen CC, Chen SC. The impact of number of drugs prescribed on the risk of potentially inappropriate medication among outpatient older adults with chronic diseases. QJM. 2013 Nov;106(11):1009-15. doi: 10.1093/qjmed/hct141. Epub 2013 Jul 8. PMID 23836694
- [Result] Fick DM, Semla TP. 2012 American Geriatrics Society Beers Criteria: new year, new criteria, new perspective. J Am Geriatr Soc. 2012 Apr;60(4):614-5. doi: 10.1111/j.1532-5415.2012.03922.x. Epub 2012 Feb 29. No abstract available. PMID 22376003
- [Result] Billioti de Gage S, Moride Y, Ducruet T, Kurth T, Verdoux H, Tournier M, Pariente A, Begaud B. Benzodiazepine use and risk of Alzheimer's disease: case-control study. BMJ. 2014 Sep 9;349:g5205. doi: 10.1136/bmj.g5205. PMID 25208536
- [Result] Kripke DF, Langer RD, Kline LE. Hypnotics' association with mortality or cancer: a matched cohort study. BMJ Open. 2012 Feb 27;2(1):e000850. doi: 10.1136/bmjopen-2012-000850. Print 2012. PMID 22371848
- [Result] Olfson M, King M, Schoenbaum M. Benzodiazepine use in the United States. JAMA Psychiatry. 2015 Feb;72(2):136-42. doi: 10.1001/jamapsychiatry.2014.1763. PMID 25517224
- [Result] Cascade E, Kalali AH. Use of benzodiazepines in the treatment of anxiety. Psychiatry (Edgmont). 2008 Sep;5(9):21-2. PMID 19727256
- [Result] Cook JM, Marshall R, Masci C, Coyne JC. Physicians' perspectives on prescribing benzodiazepines for older adults: a qualitative study. J Gen Intern Med. 2007 Mar;22(3):303-7. doi: 10.1007/s11606-006-0021-3. PMID 17356959
- [Result] Kaur S, Mitchell G, Vitetta L, Roberts MS. Interventions that can reduce inappropriate prescribing in the elderly: a systematic review. Drugs Aging. 2009;26(12):1013-28. doi: 10.2165/11318890-000000000-00000. PMID 19929029
- [Result] Crotty M, Halbert J, Rowett D, Giles L, Birks R, Williams H, Whitehead C. An outreach geriatric medication advisory service in residential aged care: a randomised controlled trial of case conferencing. Age Ageing. 2004 Nov;33(6):612-7. doi: 10.1093/ageing/afh213. Epub 2004 Sep 22. PMID 15385274
- [Result] Loganathan M, Singh S, Franklin BD, Bottle A, Majeed A. Interventions to optimise prescribing in care homes: systematic review. Age Ageing. 2011 Mar;40(2):150-62. doi: 10.1093/ageing/afq161. Epub 2011 Jan 24. PMID 21262782
- [Result] Hanlon JT, Weinberger M, Samsa GP, Schmader KE, Uttech KM, Lewis IK, Cowper PA, Landsman PB, Cohen HJ, Feussner JR. A randomized, controlled trial of a clinical pharmacist intervention to improve inappropriate prescribing in elderly outpatients with polypharmacy. Am J Med. 1996 Apr;100(4):428-37. doi: 10.1016/S0002-9343(97)89519-8. PMID 8610730
- [Result] Simon SR, Smith DH, Feldstein AC, Perrin N, Yang X, Zhou Y, Platt R, Soumerai SB. Computerized prescribing alerts and group academic detailing to reduce the use of potentially inappropriate medications in older people. J Am Geriatr Soc. 2006 Jun;54(6):963-8. doi: 10.1111/j.1532-5415.2006.00734.x. PMID 16776793
- [Result] van Eijk ME, Avorn J, Porsius AJ, de Boer A. Reducing prescribing of highly anticholinergic antidepressants for elderly people: randomised trial of group versus individual academic detailing. BMJ. 2001 Mar 17;322(7287):654-7. doi: 10.1136/bmj.322.7287.654. PMID 11250852
- [Result] Tannenbaum C, Martin P, Tamblyn R, Benedetti A, Ahmed S. Reduction of inappropriate benzodiazepine prescriptions among older adults through direct patient education: the EMPOWER cluster randomized trial. JAMA Intern Med. 2014 Jun;174(6):890-8. doi: 10.1001/jamainternmed.2014.949. PMID 24733354
- [Result] Horne R, Weinman J. Patients' beliefs about prescribed medicines and their role in adherence to treatment in chronic physical illness. J Psychosom Res. 1999 Dec;47(6):555-67. doi: 10.1016/s0022-3999(99)00057-4. PMID 10661603